CLINICAL TRIAL: NCT00095394
Title: The Efficacy and Safety of Irbesartan/HCTZ Combination Therapy as First Line Treatment for Severe Hypertension
Brief Title: Irbesartan/Hydrochlorothiazide (HCTZ) Combination Therapy as First Line Treatment for Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV131-176
Record Dates: First submitted 2004-11-03; First posted 2004-11-04 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension
Keywords: Severe Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: Irbesartan/HCTZ
- A2 (Active Comparator)
  Interventions: Drug: Irbesartan monotherapy

INTERVENTIONS:
Drug: Irbesartan/HCTZ — Tablets, Oral, Irbesartan 150mg/HCTZ 12.5 mg, Once daily, 7 weeks.
  Other Names: Avapro
  Arms: A1
Drug: Irbesartan monotherapy — Tablets, Oral, 150 mg, Once daily, 7 weeks.
  Other Names: Avapro
  Arms: A2

SUMMARY:
The purpose of this clinical research is to learn if severe hypertension can be better controlled by initially treating with a combination of drugs (Irbesartan/HCTZ), in patients who are unlikely to achieve blood pressure (B/P) control with only one drug. In addition, the study will also evaluate the safety and tolerability of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 and older;
* Willing to provide written informed consent;
* Must have uncontrolled hypertension defined as: currently untreated with a diastolic blood pressure greater than 110 mmHg OR currently receiving antihypertensive monotherapy with a diastolic blood pressure greater than 100 mmHg. Monotherapy is defined as treatment with one antihypertensive medication for at least four weeks; fixed combination therapy does not represent monotherapy;
* Must be willing to discontinue antihypertensive medication, if applicable;
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to one week after the study in such a manner that the risk of pregnancy is minimized.
* WOCBP must have a negative serum or urine pregnancy test within 72 hours prior to the start of study medication.

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Known or suspected secondary hypertension;
* Hypertension emergencies or stroke within the past 12 months;
* Heart attack, angina or bypass surgery within the past 6 months;
* Significant kidney disease;
* Significant liver disease;
* Systemic lupus erythematosus;
* Gastrointestinal disease or surgery that may interfere with drug absorption;
* Cancer during the past five years excluding localized squamous cell or basal cell carcinoma of the skin;
* Currently pregnant or lactating;
* Mental condition (psychiatric or organic cerebral disease) rendering the subject unable to understand the nature, scope, and possible consequences of the study;
* Drug or alcohol abuse within the last five years;
* Known allergy to irbesartan or diuretics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Estimated)
Dates: Start 2004-09; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects whose seated diastolic blood pressure is controlled (SeDBP < 90 mmHg) at Week 5

SECONDARY OUTCOMES:
Frequency of discontinuation due to AE, frequencies of hypotension, dizziness, syncope, headaches, hypokalemia and hyperkalemia after 17 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (269):
- United States (156):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Columbiana, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Sherwood, Arkansas
  - Local Institution, Carlsbad, California
  - Local Institution, Carmichael, California
  - Local Institution, Corona, California
  - Local Institution, Encinitas, California
  - Local Institution, Fresno, California
  - Local Institution, Laguna Hills, California
  - Local Institution, Long Beach, California
  - Local Institution, Mission Hills, California
  - Local Institution, Raleigh, California
  - Local Institution, Redondo Beach, California
  - Local Institution, Rolling Hills Estate, California
  - Local Institution, Roseville, California
  - Local Institution, Sacramento, California
  - Local Institution, San Diego, California
  - Local Institution, San Jose, California
  - Local Institution, Santa Ana, California
  - Local Institution, Torrance, California
  - Local Institution, Tustin, California
  - Local Institution, Boulder, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Highlands Ranch, Colorado
  - Local Institution, Wheat Ridge, Colorado
  - Local Institution, Bridgeport, Connecticut
  - Local Institution, Waterbury, Connecticut
  - Local Institution, Newark, Delaware
  - Local Institution, Charlotte Harbour, Florida
  - Local Institution, Chipley, Florida
  - Local Institution, Clearwater, Florida
  - Local Institution, Cocoa Beach, Florida
  - Local Institution, Crestview, Florida
  - Local Institution, DeLand, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Niceville, Florida
  - Local Institution, North Miami Beach, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, Ocoee, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Port Orange, Florida
  - Local Institution, Saint Cloud, Florida
  - Local Institution, Sarasota, Florida
  - Local Institution, Tamarac, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Vero Beach, Florida
  - Local Institution, Zephyrhills, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Peoria, Illinois
  - Local Institution, Vernon Hills, Illinois
  - Local Institution, Des Moines, Iowa
  - Local Institution, Kansas City, Kansas
  - Local Institution, Wichita, Kansas
  - Local Institution, Erlanger, Kentucky
  - Local Institution, Richmond, Kentucky
  - Local Institution, Chalmette, Louisiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Elkton, Maryland
  - Local Institution, Oxon Hill, Maryland
  - Local Institution, Ayer, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Sudbury, Massachusetts
  - Local Institution, Livonia, Michigan
  - Local Institution, Saginaw, Michigan
  - Local Institution, Cleveland, Mississippi
  - Local Institution, Olive Branch, Mississippi
  - Local Institution, Picayune, Mississippi
  - Local Institution, Manchester, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Butte, Montana
  - Local Institution, Missoula, Montana
  - Local Institution, Omaha, Nebraska
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Dover, New Hampshire
  - Local Institution, Hillsborough, New Jersey
  - Local Institution, South Bound Brook, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Buffalo, New York
  - Local Institution, East Syracuse, New York
  - Local Institution, Fulton, New York
  - Local Institution, Lake Success, New York
  - Local Institution, Mount Vernon, New York
  - Local Institution, New York, New York
  - Local Institution, Olean, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Gastonia, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, High Point, North Carolina
  - Local Institution, Mint Hill, North Carolina
  - Local Institution, Nashville, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Canton, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Genoa, Ohio
  - Local Institution, Kettering, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Perrysburg, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Eugene, Oregon
  - Local Institution, Medford, Oregon
  - Local Institution, Orangeburg, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Bensalem, Pennsylvania
  - Local Institution, Camp Hill, Pennsylvania
  - Local Institution, Collegeville, Pennsylvania
  - Local Institution, Levittown, Pennsylvania
  - Local Institution, Penndel, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, West Grove, Pennsylvania
  - Local Institution, Cranston, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Columbia, South Carolina
  - Local Institution, Landrum, South Carolina
  - Local Institution, Prosperity, South Carolina
  - Local Institution, Saluda, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Summerville, South Carolina
  - Local Institution, Bartlett, Tennessee
  - Local Institution, Bristol, Tennessee
  - Local Institution, Cordova, Tennessee
  - Local Institution, Hendersonville, Tennessee
  - Local Institution, Johnson City, Tennessee
  - Local Institution, Morristown, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, New Tazewell, Tennessee
  - Local Institution, Selmer, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Colleyville, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Lake Jackson, Texas
  - Local Institution, Midland, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, The Colony, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Burke, Virginia
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Hampton, Virginia
  - Local Institution, Norfolk, Virginia
  - Local Institution, Lacey, Washington
  - Local Institution, Olympia, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Madison, Wisconsin
  - Local Institution, Milwaukee, Wisconsin
- Belgium (10):
  - Local Institution, Huy, Luik
  - Local Institution, Antwerp
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Genk
  - Local Institution, Hasselt
  - Local Institution, La Louvière
  - Local Institution, Liège
  - Local Institution, Roeselare
  - Local Institution, Wilrijk
- Canada (32):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Red Deer, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, North Vancouver, British Columbia
  - Local Institution, Quesnel, British Columbia
  - Local Institution, Sidney, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Aylmer, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Markham, Ontario
  - Local Institution, Niagra Falls, Ontario
  - Local Institution, Oakville, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Richmond Hill, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Montague, Prince Edward Island
  - Local Institution, Bonaventure, Quebec
  - Local Institution, Chandler, Quebec
  - Local Institution, Chicoutimi, Quebec
  - Local Institution, Drummondville, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- France (21):
  - Local Institution, Ambrières-les-Vallées
  - Local Institution, Angers
  - Local Institution, Bagneux
  - Local Institution, Bouère
  - Local Institution, Château-Gontier
  - Local Institution, Cherbourg
  - Local Institution, Équeurdreville-Hainneville
  - Local Institution, Évron
  - Local Institution, La Glacerie
  - Local Institution, La Rochelle
  - Local Institution, Laval
  - Local Institution, Le Lion-dAngers
  - Local Institution, Longue
  - Local Institution, Longué-Jumelles
  - Local Institution, Louverné
  - Local Institution, Mayenne
  - Local Institution, Nieul-sur-Mer
  - Local Institution, Noyant
  - Local Institution, Sainte-Suzanne
  - Local Institution, Saumur
  - Local Institution, Villebernier
- Germany (27):
  - Local Institution, Spaichingen, Baden-Wurttembe
  - Local Institution, Loxstedt, Niedersach
  - Local Institution, Beckum
  - Local Institution, Berlin
  - Local Institution, Blankenhain
  - Local Institution, Essen
  - Local Institution, Flörsheim
  - Local Institution, Frankfurt
  - Local Institution, Fürth
  - Local Institution, Georgsmarienhütte
  - Local Institution, Germersheim
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Krombach
  - Local Institution, Künzing
  - Local Institution, Lambrecht
  - Local Institution, Mainburg
  - Local Institution, Mannheim
  - Local Institution, Messkirch
  - Local Institution, Monheim
  - Local Institution, Nuremberg
  - Local Institution, Parsberg
  - Local Institution, Pforzheim
  - Local Institution, Stuttgart
  - Local Institution, Villingen-Schwenningen
  - Local Institution, Waldbrunn
  - Local Institution, Welver
- Israel (8):
  - Local Institution, Beersheba
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Matan
  - Local Institution, Tel Litwinsky
  - Local Institution, Ẕerifin
- Netherlands (12):
  - Local Institution, Beek en Donk
  - Local Institution, Eindhoven
  - Local Institution, Hardenberg
  - Local Institution, Heerlen
  - Local Institution, Lichtenvoorde
  - Local Institution, Rijswyk Zh
  - Local Institution, The Hague
  - Local Institution, Tilburg
  - Local Institution, Venlo
  - Local Institution, Waalwijk
  - Local Institution, Woerden
  - Local Institution, Zeist
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov